CLINICAL TRIAL: NCT06439433
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Phase IIc Clinical Trial of ALA-PDT in Patients With Cervical Intraepithelial Neoplasia Grade 2 (CIN2) in p16-positivity and High-risk HPV Infection
Brief Title: ALA-PDT in Patients With CIN2 in p16-positivity and High-risk HPV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FDZJYX-ALA-202001
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Cervical Intraepithelial Neoplasia Grade 2; Papillomavirus Infections; p16 Protein
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ALA A Group (Experimental): ALA 500mg Group
  Interventions: Drug: Aminolaevulinic acid (500-mg bottle)
- ALA B Group (Experimental): ALA 750mg Group
  Interventions: Drug: Aminolaevulinic acid (750-mg bottle)
- Placebo (Placebo Comparator): Placebo Group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aminolaevulinic acid (500-mg bottle) — once a week for 6 weeks
  Other Names: ALA 500mg
  Arms: ALA A Group
Drug: Aminolaevulinic acid (750-mg bottle) — once a week for 6 weeks
  Other Names: ALA 750mg
  Arms: ALA B Group
Drug: Placebo — once a week for 6 weeks
  Arms: Placebo

SUMMARY:
Efficacy and Safety of ALA-PDT in patients with cervical intraepithelial neoplasia grade 2 (CIN2) in p16-positivity and high-risk HPV infection.

DETAILED DESCRIPTION:
A multi-center, randomized, double-blind, placebo-controlled phase IIc clinical trial of ALA-PDT in patients with cervical intraepithelial neoplasia grade 2 (CIN2) in p16-positivity and high-risk HPV infection.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women, 18-45 years of age
* Satisfactory the colposcopy examination (cervical transformation zone types: Type 1 or 2) at screening, and CIN2 as verified by cervical biopsy and p16-positivity within the last 3 months
* Intense desire to retain the cervical structure or function
* High-risk (including probably/possibly carcinogenic) HPV-DNA (i.e. 16, 18, 26, 31, 33, 35, 39, 45, 51, 52, 53, 56, 58, 59, 66, 68, 73 or 82) positive within the last 3 months
* Meet the following conditions: pregnancy test negative; no pregnancy plan during the trial;no sexuality or reliable contraceptive measures taken since last menstruation to the onset of the study, agreeing to adopt reliable contraceptive measures during the study
* Signed written informed consent

Exclusion Criteria:

* Atypical glandular cells (AGS) or adenocarcinoma in situ (AIS) on cytology ,or malignant cells on cytology or histology, or other suspicion of either micro-invasive or invasive disease
* Invasive carcinoma possibility or lesions extending to the vaginal wall
* Severe pelvic inflammatory disease, severe cervicitis, or other severe gynaecological infection as per clinical examination
* Undiagnosed vaginal bleeding within the last 3 months
* With allergic disease at present; known or suspected porphyria; known allergy to ALA or analogues
* With serious cardiovascular, neurologic, psychiatric, endocrine, hematological disease; immunocompromised conditions or long-term glucocorticoid or immunosuppressants exposure; patients with malignant tumors within the last 5 years
* Hepatic or renal functions abnormal (alanine aminotransferase or aspartate transaminase > 3 upper limit of normal [ULN], or total bilirubin > 1.5 ULN, or serum creatinine or blood urea nitrogen > 1.5 ULN)
* History of treatment with systemic antivirals (continued for ≥ 14 days) within the last 3 months
* Pregnancy or nursing
* Participation in any clinical studies within the last 30 days
* Poor compliance or inability to complete the trial
* Subjects that the investigators judged to be not suitable to participate the study besides above

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
Response rate at week 12 after last treatment | Baseline and week 12 after treatments
  "Response" is defined as: pathology showed normal or only inflammatory changes or CIN1

SECONDARY OUTCOMES:
Response rate at week 24 after last treatment | Baseline and week 24 after treatments
  "Response" is defined as: pathology showed normal or only inflammatory changes or CIN1
Cure rate at week 12 after last treatment | Baseline and week 12 after treatments
  "Cure" is defined as: pathology showed normal or only inflammatory changes
Cure response rate at week 24 after last treatment | Baseline and week 24 after treatments
  "Cure" is defined as: pathology showed normal or only inflammatory changes
Clearance rate of HPV at week 12 after last treatment | Baseline and week 12 after treatments
  Proportion of patients with HPV clearance
Clearance rate of HPV at week 24 after last treatment | Baseline and week 24 after treatments
  Proportion of patients with HPV clearance

OTHER OUTCOMES:
Response rate of HPV16 and/or HPV18 positive patients at week 12 after last treatment | Baseline and week 12 after treatments
  "Response" is defined as: pathology showed normal or only inflammatory changes or CIN1
Response rate of HPV16 and/or HPV18 positive patients at week 24 after last treatment | Baseline and week 24 after treatments
  "Response" is defined as: pathology showed normal or only inflammatory changes or CIN1

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The Obstetrics & Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Renji Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality